CLINICAL TRIAL: NCT02229292
Title: Prevention of Bleeding and Edema in Bimaxillary Orthognathic Surgery; the Effectiveness of Tranexamic Acid on Intraoperative Bleeding and Postoperative Swelling in Orthognathic Surgery.
Brief Title: Prevention of Intraoperative Bleeding and Postoperative Swelling in Orthognathic Surgery Through the Use of Tranexamic Acid
Acronym: TXA2014-15
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: University of Copenhagen (Other); Vestjydsk Ortopædisk Fond (Unknown)
Responsible Party: Principal Investigator, Jesper Jared Olsen, DDS, Esbjerg Hospital - University Hospital of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2013-005473-52
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Intraoperative Bleeding; Postoperative Edema
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic acid (Active Comparator): The active comparator consists of an intravenously administered bolus injection of 10ml of 100mg/ml tranexamic (1g in total) given as a single dose, after the onset of anesthesia, prior to surgery.
  Interventions: Drug: Tranexamic Acid
- Saline (Placebo Comparator): The placebo consists of an intravenously administered bolus injection of 10 ml of 9mg/ml sodium chloride given as a single dose after the onset of anesthesia, prior to surgery.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Tranexamic Acid — Active group:
  Undergoes elective bi-maxillary orthognathic surgery consisting of a (un)/segmented LeFort I osteotomy combined with a bilateral sagittal split osteotomy, under the influence of 10ml tranexamic acid (100mg/ml) administered iv. prior to the onset of the surgical procedure.
  Other Names: Tranexamsyre "Pfizer", D.SP.NR.: 22646, ATC code: B 02 AA 02
  Arms: Tranexamic acid
Drug: Saline — Placebo group:
  Undergoes elective bi-maxillary orthognathic surgery consisting of a (un)/segmented LeFort I osteotomy combined with a bilateral sagittal split osteotomy, under the influence of 10ml sodium chloride (9mg/ml) administered iv. prior to the onset of the surgical procedure.
  Other Names: Natriumklorid "B. Braun", D.SP.NR.: 6856, ATC code: V 07 AB
  Arms: Saline

SUMMARY:
Purpose of the study:

* To evaluate the effect of tranexamic acid (TXA) of intraoperative blood loss in patients subjected to bi-maxillary orthognathic surgery
* To evaluate the potential effect of TXA on fibrin structure
* To evaluate the potential effect of TXA of binding of plasminogen to fibrin
* To evaluate the potential effect of TXA on postoperative edema formation.

Hypothesis:

H0: Intraoperative bleeding cannot be significantly reduced by preoperative administration of tranexamic acid

H0,1: Postoperative edema cannot be significantly reduced by preoperative administration of tranexamic acid

DETAILED DESCRIPTION:
The study population consists of patients referred to simultaneous mandibular and maxillary osteotomy at the Department of Oral and Maxillofacial Surgery, Hospital of South West Denmark in 2014.

Hundred patients (50 men and 50 women) will be enrolled in the study. Reportedly, the mean intraoperative blood loss in the placebo group is expected to be 436 ml with a standard deviation of 208 ml. The difference in blood loss between the TXA-group and the placebo group to be detected is 100 ml. The dropout frequency is estimated to 10%. To fulfil these assumptions a minimum of 40 patients should be included in each group to reach a power of 0.8 and an alpha of 0.05. In order to accommodate an even gender distribution a block randomization is performed resulting in the randomization of 100 patients.

The patients will be randomized to receive blindly either 10 ml tranexamic acid (100 mg/ml) (Pfizer, Ballerup, Denmark) or 10 ml saline (9mg/ml) preoperatively. Intraoperative blood loss will be determined by deducting the total volume of irrigation fluids from the volume of the contents of the surgical suction device. Postoperative edema formation will be determined by 3D surface scanning and volumetric analysis will be carried out in the "Landmarker" software.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older
* Patients must be eligible for elective bi-maxillary orthognathic surgery
* No severe reduction of kidney function
* No known medical conditions
* Signed informed consent

Exclusion Criteria:

* Hypersensitivity to tranexamic acid
* A medical history of acute venous thrombosis and/or arterial thrombosis
* The presence of fibrinolytic conditions as a result of disseminated intravascular coagulation, with the exception of a predominant activation of the fibrinolytic system with acute severe bleeding.
* Severe kidney deficiency
* Cramps in the medical history
* Intake of Omega-3 fatty acids, Gingko Biloba, ginger and garlic supplements within 3 months of surgery.
* Pregnancy (female participants will be tested on the day of surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-08-19; Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-26 (Actual)

PRIMARY OUTCOMES:
Intra-operative bleeding volume (ml) | Within 10 minutes after ended surgery

SECONDARY OUTCOMES:
Change in hemostatic profile | Baseline, 5.5 hours, 48 hours and 4 months postoperatively
  Changes in the hemostatic profile measured through thrombelastography, thrombin generation test and fibrin structure analysis.
Change in inflammatory profile | Baseline, 5.5 hours, 48 hours and 4 months postoperatively
  Changes in the inflammatory profile are investigated through measures of surface induced activation, inflammation and plasminogen binding.
Postoperative edema formation | 48 hours and 4 months postoperatively
  The degree of postoperative swelling in connection with TXA /or not, is determined by non-invasive 3D face scans and quantified using the "Landmarker" software. Scans are carried out along with the 3rd and 4th blood samples, 48 hours and 4 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper J Olsen, DDS, Principal Investigator — Esbjerg Hospital - University Hospital of Southern Denmark
Locations (1):
- Hospital of South West Denmark, Esbjerg, Denmark

REFERENCES:
- [Background] Song G, Yang P, Hu J, Zhu S, Li Y, Wang Q. The effect of tranexamic acid on blood loss in orthognathic surgery: a meta-analysis of randomized controlled trials. Oral Surg Oral Med Oral Pathol Oral Radiol. 2013 May;115(5):595-600. doi: 10.1016/j.oooo.2012.09.085. Epub 2012 Dec 20. PMID 23260768